CLINICAL TRIAL: NCT00974805
Title: An Investigation Into the Mechanisms of Action of a Combined Long Acting Beta Agonist/Inhaled Corticosteroid (Seretide 500 Accuhaler) on the Bacterial Colonisation, Immunology and Inflammation of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: An Investigation of the Mechanism of Action of Seretide in Chronic Obstructive Pulmonary Disease
Acronym: IMAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SCB-001
Record Dates: First submitted 2009-09-08; First posted 2009-09-10 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Emphysema; Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Seretide 500 Accuhaler (Experimental): Seretide 500 Accuhaler one inhalation BD
  Interventions: Drug: Seretide 500 Accuhaler

INTERVENTIONS:
Drug: Seretide 500 Accuhaler — Seretide 500 accuhaler one inhalation BD

SUMMARY:
This study is investigating the possible mechanisms of action of an inhaled treatment (Seretide), currently used worldwide in millions of patients with COPD (Chronic Obstructive Pulmonary Disease) and how it improves the symptoms of these patients. Previous research has failed to identify the mechanisms at play other than dilation of the airways. The research community has long thought the mechanism to be immune based or anti inflammatory but despite intensive research this has not yet been identified.

DETAILED DESCRIPTION:
We aim to recruit equal numbers of healthy smokers, mild, moderate and severe COPD patients (12 patients to be recruited from each group). These patients will never have been prescribed the components present in Seretide (Salmeterol and Flixotide or similar compounds).

The patients will have spirometry at the beginning of the study to confirm the presence of COPD. Healthy smokers will defined as ex or current smokers who match the study population but have normal lung function.

Patients with a history of asthma, bronchiectasis, carcinoma of the bronchus, or other significant respiratory disease will be excluded.

The patients will have a total of four study visits, 2 off treatment and 2 while on treatment, over a 56 day study period. At each study visit induced sputum will be performed and blood extracted. The cells fom both of these samples will be analysed for cells type and activation. Sputum and serum will be stored for cytokine analysis at a later date.

The Sputum will be induced using standardised protocols using nebulised saline solution.

ELIGIBILITY:
Inclusion Criteria:

* >35yrs.
* >10 Pack Years COPD as defined as an FEV1<70% and an FEV1/FVC ratio of <70%

Exclusion Criteria:

* Asthma
* Lung cancer
* Bronchiectasis

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are change in cell type and activation status | 56 days

SECONDARY OUTCOMES:
Change in sputum and serum cytokines Change in bacterial colonization | 56 days

CONTACTS AND LOCATIONS:
Locations (1):
- Southampton General Hospital, Southampton, Hampshire, United Kingdom